CLINICAL TRIAL: NCT06390722
Title: A Phase 3b/4 Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Effect of Upadacitinib on Atopic Dermatitis-induced Sleep Disturbance in Adults With Moderate to Severe Atopic Dermatitis (SLEEP UP)
Brief Title: A Study to Assess the Effect of Upadacitinib in Atopic Dermatitis-induced Sleep Disturbance in Adults With Moderate to Severe Atopic Dermatitis
Acronym: Sleep Up
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: strategic decision
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: M24-602
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Atopic Dermatitis; Sleep Disturbance
Keywords: Upadacitinib; RINVOQ; ABT-494; Atopic Dermatitis; Sleep Disturbance
MeSH Terms: conditions — Dermatitis, Atopic; Parasomnias | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Upadacitinib (Experimental): Participants randomized to receive upadacitinib Dose A once daily for 2 weeks during double-blind treatment period. At week 2, participants will be switched to open-label upadacitinib Dose A once daily for 22 weeks.
  Interventions: Drug: Upadacitinib
- Placebo (Placebo Comparator): Participants randomized to receive Placebo once daily for 2 weeks during double-blind treatment period. At week 2, participants will be switched to open-label upadacitinib Dose A once daily for 22 weeks.
  Interventions: Drug: Placebo for Upadacitinib

INTERVENTIONS:
Drug: Upadacitinib — Oral Tablet
  Other Names: RINVOQ
  Arms: Upadacitinib
Drug: Placebo for Upadacitinib — Oral Tablet
  Arms: Placebo

SUMMARY:
Many people with atopic dermatitis (AD) experience sleep disturbances. Greater sleep disturbances are associated with greater burden including increased sick days and impaired cognition. Patient focused research has found that sleep was one of the 3 most problematic symptoms for people with AD and their families.

Upadacitinib demonstrated clinically meaningful sleep improvement based on patient-reported outcome measures such as the Atopic Dermatitis Impact Scale (ADerm-IS) Sleep Domain score in Phase 3 registrational trials, but objective data on upadacitinib's effect on elements of sleep disturbance such as Wake After Sleep Onset, or Sleep Efficiency, have not been collected.

Upadacitinib is an approved drug for the treatment of moderate to severe atopic dermatitis (AD). This study is conducted in 2 Periods. During Period 1, participants are randomly assigned into 1 of 2 groups called treatment arms to receive upadacitinib or Placebo. In Period 2, participants will be switched to receive open-label upadacitnib. Approximately 112 adult participants ages 25 to 63 with moderate to severe AD who have moderate to severe sleep disturbance will be enrolled at up to 32 sites worldwide.

This study consists of a 35-day Screening Period; a 2-week randomized, double-blinded period (Period 1); a 22-week open-label extension period (Period 2); and a 30-day follow-up visit/call. Participants will receive oral tablets once per day of Upadacitinib or Placebo for 2 weeks followed by Upadacitinib oral tablet for 22 weeks

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* AD, according to Hanifin and Rajka criteria, with onset of symptoms at least 3 years prior to Baseline.
* Eczema Area and Severity Index (EASI) score >= 16; validated Investigator Global Assessment scale for Atopic Dermatitis (vIGA-AD) score >= 3, and >= 10% Body Surface Area (BSA) of AD involvement at the Baseline Visit.
* Baseline weekly average of daily Worst Pruritus Numeric Rating Scale (NRS) >= 7.
* Moderate to severe sleep disturbance as confirmed by Baseline Patient Global Impression (PGI) Sleep AD (7-day) score of 3 or 4.
* Documented history of inadequate response to at least 1 prior systemic treatment for AD OR for whom systemic treatments, other than upadacitinib, are medically inadvisable (e.g., because of important side effects or safety risks).

Exclusion Criteria:

* Prior exposure to dupilumab, tralokinumab, lebrikizumab, or nemolizumab.
* Conditions or circumstances that could interfere with sleep assessments, including but not limited to:

  * History of sleep apnea, hypersomnia, or insomnia related to chronic pain;
  * Participant uses a continuous positive airway pressure (CPAP) machine;
  * History of chronic obstructive pulmonary disease or uncontrolled asthma;
  * Evidence of restless leg syndrome;
  * Participant is an evening or night shift worker;
  * Participant has sleep disturbance due to menopause, nocturia, or situational circumstances (e.g., caring for infant).
* Participants who had prior exposure to any oral JAK inhibitor

Ages: 25 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-05-23 (Estimated); Primary Completion 2026-01-05 (Estimated); Study Completion 2026-07-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants achieving an improvement (reduction) in Worst Pruritus Numeric Rating Scale ≥ 4 from Baseline | Baseline to Week 2
  The Worst Pruritus Numeric Rating Scale is an assessment tool that participants used to report the intensity of their pruritus during a daily recall period. On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst imaginable itch'.

SECONDARY OUTCOMES:
Change from Baseline in Total Scratch Time | Baseline to Week 2
  Scratch time will be measured in duration of seconds based on a wearable scratch sensor per sleep opportunity hour at Week 2 .
  Note: Sleep opportunity is defined as total time spent trying to sleep [i.e., sleep sensor on to sensor off time].
Change from Baseline in Sleep Efficiency | Baseline to Week 2
  A wearable sleep sensor collects actigraphy, temperature, and heart rate data to quantify sleep parameters
Change from Baseline in Wake After Sleep Onset (WASO) based on a sleep sensor. | Baseline to Week 2
  A wearable sleep sensor collects actigraphy, temperature, and heart rate data to quantify sleep parameters
Change from Baseline in Nocturnal Scratching Bouts (≥ 5 seconds) | Baseline to Week 2
  Scratch time will be measured in duration of seconds based on a wearable scratch sensor per sleep opportunity hour at Week 2 .
  Note: Sleep opportunity is defined as total time spent trying to sleep [i.e., sleep sensor on to sensor off time].

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-602